CLINICAL TRIAL: NCT04232267
Title: Development and Validation of an Algorithm to Identify a Clinically Significant Depressive Burden in Individuals Referred to Sleep Clinics for Polysomnography (PSG) Assessment (Sleep Analysis of Depressive Burden - SADB)
Brief Title: Analysis of Sleep Study Data to Assess Depressive Burden
Acronym: SADB
Status: Completed | Type: Observational
Sponsor: Medibio Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-0018
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Sleep Disorder; Depressive; Behavioral Disorder; Mood Disorders
MeSH Terms: conditions — Sleep Wake Disorders; Mental Disorders; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients prescribed Polysomnology (PSG - sleep study): Patients that are at least 18 years old but not older than 75 years old, who have been referred to a sleep clinic for sleep disturbance.
  Interventions: Device: MEB-001

INTERVENTIONS:
Device: MEB-001 — Software medical device used to aid in the screening of patients with potential depressive burden symptoms.

SUMMARY:
This study evaluates the effectiveness of the MEB-001 device in assessing physiological parameters that provide a clinically significant depressive burden screener. This study uses objective physiological markers from MEB-001 to estimate the clinically significant depressive burden as subjectively reported by the subject with the Beck Depression Inventory - II (BDI-II).

DETAILED DESCRIPTION:
This study evaluates the effectiveness of the MEB-001 device in assessing physiological parameters that provide a clinically significant depressive burden screener. This study uses objective physiological markers from MEB-001 to estimate the clinically significant depressive burden as subjectively reported by the subject with the BDI-II.

This is a two (2)-phase, non-significant risk, cross-sectional, naturalistic, single-arm, multi-center study conducted under a common protocol and designed to:

Phase 1: MEB-001 algorithm development (software medical device). Phase 2: Evaluate the effectiveness of the MEB-001 device in assessing physiological parameters that provide clinically significant depressive burden screener.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age ≥18 years and ≤75 years.
* Subject is willing and able to provide consent.
* Subject has the ability to read and understand the instructions for the study.
* Subject is willing to adhere to study procedures.
* Subject is willing to undergo full night PSG study, as prescribed.

Exclusion Criteria:

* Subject has a pacemaker.
* Subject is suspected or known to have active alcohol or drug abuse (including but not limited to abuse of marijuana).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are at least 18 years old but not older than 75 years old, who have been referred to a sleep clinic for sleep disturbances and sign an informed consent form (ICF) will be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Report assists in the detection of clinically significant depressive burden. | The study consists of 1 study visit (baseline).
  Utilize PSG data and BDI-II to determine clinical depressive burden.
Evaluate algorithm accuracy, sensitivity and specificity. | The study consists of 1 study visit (baseline).
  Sensitivity: True Positive/BDI-II + (the percentage of BDI-II positives identified by MEB-001) Specificity: True Negative/BDI-II - (the percentage of BDI-II negatives identified by MEB-001)

SECONDARY OUTCOMES:
Evaluate positive predictive value and negative predictive value in detecting clinically significant depressive burden. | The study consists of 1 study visit (baseline).
  Positive predictive value: True Positive/MEB-001 + (the percentage of MEB-001 positive test results that agree with BDI-II) Negative predictive value: True Negative/MEB-001 - (the percentage of MEB-001 negative test results that agree with BDI-II)
System reliability and internal consistency. | The study consists of 1 study visit (baseline).
  The MEB-001 is able to assess clinically depressive burden compared to the BDI-II

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bruner, Study Director — Medibio Limited; Archie Defillo, MD, Study Chair — Medibio Limited; Archie Defillo, MD, Principal Investigator — Medibio Limited
Locations (5):
- United States (5):
  - Restore Sleep Clinic, Blaine, Minnesota
  - Lakeland Sleep and CPAP, Plymouth, Minnesota
  - Ohio Sleep Solutions, Columbus, Ohio
  - Ohio Sleep Solutions, Grove City, Ohio
  - Ohio Sleep Solutions, Hilliard, Ohio

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the participant data to other researchers.